CLINICAL TRIAL: NCT02747771
Title: The Norwegian Trichotillomania Project
Brief Title: Cognitive Behavioral Group Therapy for Trichotillomania (Hair Pulling Disorder)
Acronym: NorTriP
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Sorlandet Hospital HF (Other Government); St. Olavs Hospital (Other); Texas A&M University (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Benjamin Hummelen, MD, PhD, Oslo University Hospital
Other Study IDs: 2013/632
Record Dates: First submitted 2016-04-14; First posted 2016-04-22 (Estimated); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Trichotillomania
Keywords: effectiveness; trichotillomania; hair pulling; habit reversal training; acceptance and commitment therapy; cognitive behavioral therapy
MeSH Terms: conditions — Trichotillomania | interventions — Cognitive Behavioral Therapy; Acceptance and Commitment Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — 10 sessions Group therapy during 10-12 weeks. The first three sessions focus on habit reversal training, the fourth to sixth session on acceptance and commitment therapy and the last four sessions aims at integrating the two approaches.
  Other Names: Acceptance and commitment therapy (ACT); Habit reversal training (HRT)

SUMMARY:
This study aims at evaluating the effectiveness of group-based cognitive behavioral therapy for trichotillomania at three clinical sites in Norway.

DETAILED DESCRIPTION:
The Norwegian Trichotillomania Project is a multicenter study that aims at evaluating the effectiveness of behavioral group therapy for TTM, i.e., ACT (Acceptance and commitment therapy) enhanced habit reversal training (ACT-enhanced HRT).

Participants are adults or adolescents (16 year or older) who fulfill criteria for TTM according to DSM-IV. Inclusion started in January 2013 and will be completed by Mai 2016. Treatment is delivered at three treatment sites in Norway; in Kristiansand, Oslo, and Trondheim. Treatment is manualized, following the manual of Twohig and Woods, and consists of ten group sessions of three hours delivered at consecutive weeks, and two or three booster sessions during the first year after treatment.

Treatment outcome is evaluated by three outcome measures; the Massachusetts General Hospital - Hairpulling Scale (self-report); the National Institute of Mental Health Trichotillomania Severity Scale (clinical interview, conducted by independent evaluators); and the Clinical Global Impression Scale for TTM. Outcome is measured at three points in time; at baseline, at the end of treatment, and at one-year follow-up. Mixed models procedures in SPSS is used to analyze longitudinal data.

The first paper will be written on patients admitted to treatment from January 2013 to September 2014, and includes 53 patients (49 women and four men). By January 2016, fifty-one patients (96%) had participated in the one-year follow-up evaluation.

ELIGIBILITY:
* Inclusion Criteria:

  * Clinical diagnosis of Trichotillomania
  * Age between 16 and 67
* Exclusion Criteria:

  * schizophrenia spectrum disorder
  * substance addiction
  * severe antisocial, schizotypal, or paranoid personality disorder
  * severe eating disorder,
  * ongoing suicidal ideation
  * pervasive developmental disorder
  * mental retardation and severe sequelae after brain injury.

Ages: 16 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred for treatment of trichotillomania (TTM)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-01-01; Primary Completion 2024-04-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in National Institute of Mental Health Trichotillomania Severity Scale (NIMH-TSS) | baseline, 12 weeks, 12 months
  clinical interview
Change in Massachusetts General Hospital - Hairpulling Scale (MGH-HS) | baseline, 12 weeks, 12 months
  self-report

SECONDARY OUTCOMES:
Change Patient Health Questionnaire-9 (PHQ-9) | baseline, 12 weeks, 12 months
  self-report depressive symptoms
Change General Anxiety Disorder Scale (GAD-7) | baseline, 12 weeks, 12 months
  self-report anxiety symptoms
Change Metacognition Questionnaire (MCQ-30) | baseline, 12 weeks, 12 months
  self-reported metacognitions
Change in Acceptance and Action Questionnaire for Trichotillomania | baseline, 12 weeks, 12 months
  self-report

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Hummelen, Ph.D., M.D., Principal Investigator — Oslo University Hospital, Oslo, Norway
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stein DJ, Grant JE, Franklin ME, Keuthen N, Lochner C, Singer HS, Woods DW. Trichotillomania (hair pulling disorder), skin picking disorder, and stereotypic movement disorder: toward DSM-V. Depress Anxiety. 2010 Jun;27(6):611-26. doi: 10.1002/da.20700. PMID 20533371
- [Background] Stein DJ, Garner JP, Keuthen NJ, Franklin ME, Walkup JT, Woods DW. Trichotillomania, stereotypic movement disorder, and related disorders. Curr Psychiatry Rep. 2007 Aug;9(4):301-2. doi: 10.1007/s11920-007-0036-4. PMID 17880861
- [Background] Woods DW, Wetterneck CT, Flessner CA. A controlled evaluation of acceptance and commitment therapy plus habit reversal for trichotillomania. Behav Res Ther. 2006 May;44(5):639-56. doi: 10.1016/j.brat.2005.05.006. Epub 2005 Jul 22. PMID 16039603
- [Background] Keuthen NJ, Rothbaum BO, Fama J, Altenburger E, Falkenstein MJ, Sprich SE, Kearns M, Meunier S, Jenike MA, Welch SS. DBT-enhanced cognitive-behavioral treatment for trichotillomania: A randomized controlled trial. J Behav Addict. 2012 Sep;1(3):106-14. doi: 10.1556/JBA.1.2012.003. PMID 26165460
- [Result] Houghton DC, Capriotti MR, De Nadai AS, Compton SN, Twohig MP, Neal-Barnett AM, Saunders SM, Franklin ME, Woods DW. Defining treatment response in trichotillomania: a signal detection analysis. J Anxiety Disord. 2015 Dec;36:44-51. doi: 10.1016/j.janxdis.2015.09.008. Epub 2015 Sep 24. PMID 26422605